CLINICAL TRIAL: NCT03503682
Title: SHort Course Accelerated RadiatiON Therapy (SHARON) in Complicated Bone Metastases Palliation: an Interventional, Randomised, Multicentric Study
Brief Title: Short Course Radiation Therapy in Palliative Treatment of Complicated Bone Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT-15-06 SHARON BONE
Record Dates: First submitted 2018-04-09; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Bone Metastases; Radiotherapy; Palliative Care
Keywords: Short Course Radiotherapy; Complicated Bone Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard treatment (Active Comparator): Patients in this group are treated with 3000 cGy in 10 daily fractions
  Interventions: Radiation: standard treatment
- short course treatment (Experimental): Patients in this group are treated with 2000 cGy in 4 fractions administered twice a day (at least 6-8 hours interval)
  Interventions: Radiation: short course treatment

INTERVENTIONS:
Radiation: standard treatment — 3000 cGy in 10 daily fractions
  Arms: standard treatment
Radiation: short course treatment — 2000 cGy in 4 fractions administered twice a day
  Arms: short course treatment

SUMMARY:
Aim of the study is to assess efficacy of a short course radiation treatment in patients with complicated bone metastases

DETAILED DESCRIPTION:
Standard treatment for complicated bone metastases (3000 cGy in 10 daily fractions of 300 cGy each) is compared with experimental treatment (4000 cGy in 4 fractions of 500 cGy twice a day) to demonstrate non-inferiority of this scheme.

ELIGIBILITY:
Inclusion Criteria:

* complicated bone metastases from any solid tumor
* age >18 years
* ECOG performance status 0-3
* symptomatic lesion (NRS >1)
* no changes in analgesic treatment at least in the week before radiotherapy

Exclusion Criteria:

* pregnancy
* previously irradiation of the same region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2022-11-08 (Estimated); Study Completion 2023-11-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of palliation using the short course scheme compared with the standard scheme | 3 months
  Reduction of pain after radiotherapy, assessed with VAS (visual analogue scale)

SECONDARY OUTCOMES:
Acute toxicity in the two treatment groups | 3 months
  incidence of treatment-related acute adverse events in the two arms of the study registered using Cooperative Group Common Toxicity Criteria
Late toxicity in the two treatment groups | 12 months
  incidence of treatment-related late adverse events in the two arms of the study registered using RTOG/EORTC Late Radiation Morbidity Scoring Schema
Quality of Life (QoL) assessment in the two groups | 12 months
  Changes in QoL after the treatment assessed using EORTC questionnaires (QLQ-BM22 and C15-PAL)

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, MD, Principal Investigator — Radiation Oncology Center, Department of Experimental, Diagnostic and Speciality Medicine-DIMES, Unversity of Bologna, S. Orsola-Malpighi Hospital, Bologna, Italy
Locations (1):
- Radiation Oncology Center, Department of Experimental, Diagnostic and Speciality Medicine- DIMES, University of Bologna, S.Orsola-Malpighi Hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zamagni A, Siepe G, Gibertoni D, Donati CM, Cellini F, Fiorica F, Pezzulla D, Deodato F, Candoli F, Bisello S, Scirocco E, Manfrida S, Gabbani M, Cilla S, Macchia G, Morganti AG. Accelerated Radiotherapy for Complicated Bone Metastases: SHARON Bone Randomized Phase III Trial Shows Non-Inferiority Compared to Standard Palliative Fractionation (NCT03503682). Cancers (Basel). 2025 Jun 16;17(12):2000. doi: 10.3390/cancers17122000. PMID 40563650